CLINICAL TRIAL: NCT01191008
Title: Special Investigation Of Long Term Use Of Xalacom(Regulatory Post Marketing Commitment Plan)
Brief Title: Long Term Use Of Xalacom In Patients Glaucoma Or Ocular Hypertension
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A6641056
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2017-02

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Xalacom Regulatory post marketing commitment plan safety
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Xalacom

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Latan-timolol maleate fixed comb ophthalmic solution
  Interventions: Drug: Latanoprost-timolol maleate fixed combination ophthalmic solution

INTERVENTIONS:
Drug: Latanoprost-timolol maleate fixed combination ophthalmic solution — Xalacom® Combination Eye Drops depending on the Investigator prescription. Frequency and duration are according to Package Insert as follows. "One drop should be applied to the affected eye(s) once daily".
  Other Names: Xalacom

SUMMARY:
The objective of this Investigation is to evaluate the safety and efficacy of long-term treatment with Xalacom in medical practice. Also, occurrence of unknown and known adverse drug reactions (ADRs) in subjects treated with Xalacom will be monitored during the survey period, and whether an additional treatment outcome investigation and/or a post-marketing clinical study is required in the future will be determined.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Xalacom® should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered Xalacom® in order to be enrolled in the surveillance.

Exclusion Criteria:

* Patients not administered Xalacom®.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A6641056 prescribes the Xalacom® Combination Eye Drops.
Sampling Method: Probability Sample
Enrollment: 661 (Actual)
Dates: Start 2010-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6641056&StudyName=Long%20Term%20Use%20Of%20Xalacom%20In%20Patients%20Glaucoma%20Or%20Ocular%20Hypertension

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 661 participants were registered in the study. Of the 661 participants, 28 participants were excluded from the study because their case report forms were not collected. Finally, 633 participants were included in the study.
Groups:
- Latanoprost/Timolol Maleate: Participants received latanoprost/timolol maleate fixed combination eye drops into the affected eye(s) once daily for to a maximum of 104 weeks.
Period: Overall Study
Arm/Group | Latanoprost/Timolol Maleate
Started | 633
Completed | 618
Not Completed | 15
Not completed — Protocol Violation | 7
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Population: A total of 661 participants were registered in the study. 28 participants were excluded from the study because their case report forms were not collected.Of the 633 participants, 15 participants were excluded from the baseline analysis due to following reasons: protocol violation (7 participants) and lost to follow-up (8 participants).
Arm/Group | Latanoprost/Timolol Maleate
Number analyzed (Participants) | 618
Age, Customized [Number; unit: Participants]
  >=15 and <65 years | 227
  ˃=65 years | 391
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 329
  Male | 289

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants WithTreatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to latanoprost/timolol maleate in a participant who received latanoprost/timolol maleate. Relatedness to latanoprost/timolol maleate was assessed by the investigator.
Time Frame: Max 104 weeks
Population: The safety analysis set comprised of participants who had met the inclusion criteria and had received latanoprost/timolol maleate at least once.
Measure: Number; unit: Participants
Arm/Group | Latanoprost/Timolol Maleate
Number analyzed (Participants) | 618
Participants | 73

2. Primary Outcome: Clinical Effectiveness Rate
Description: Clinical effectiveness rate, which was defined as the percentage of participants who achieved clinical effectiveness over the total number of effectiveness analysis population, was presented along with the corresponding exact 2sided 95% confidence interval. Overall effectiveness of latanoprost/timolol was determined by the investigator based on clinical symptoms and examinations. Clinical effectiveness was assessed according to the following categories: (1) effective, (2) not effective, or (3) not assessable at the end of observation period (Max 104 weeks).
Time Frame: Max 104 weeks
Population: The effectiveness analysis set comprised of participants that were excluded off-label uses or blank evaluation from safety analysis set.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Latanoprost/Timolol Maleate
Number analyzed (Participants) | 618
Percentage of participants | 82.8 [79.6 to 85.7]

3. Other Pre Specified Outcome: Number of Participants With Treatment-Related Adverse Events Unexpected From Japanese Package Insert
Description: A treatment-related adverse event was any untoward medical occurrence attributed to latanoprost/timolol maleate in a participant who received latanoprost/timolol maleate. Expectedness of the adverse event was determined according to Japanese package insert. Relatedness to latanoprost/timolol maleate was assessed by the investigator.
Time Frame: Max 104 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Latanoprost/Timolol Maleate
Number analyzed (Participants) | 618
Participants | 3

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Latanoprost/Timolol Maleate
Serious Adverse Events (participants affected / at risk) | 13/618
Other Adverse Events (participants affected / at risk) | 134/618
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Latanoprost/Timolol Maleate (N=618)
Ophthalmic herpes zoster (Infections and infestations) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Marasmus (Metabolism and nutrition disorders) | 1
Age-related macular degeneration (Eye disorders) | 1
Corneal disorder (Eye disorders) | 1
Blindness (Eye disorders) | 1
Cataract (Eye disorders) | 3
Retinoschisis (Eye disorders) | 1
Angina unstable (Cardiac disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 1
Intraocular pressure increased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Latanoprost/Timolol Maleate (N=618)
Conjunctivitis (Infections and infestations) | 11
Conjunctivitis bacterial (Infections and infestations) | 1
Visual field defect (Nervous system disorders) | 2
Uveitis (Eye disorders) | 3
Conjunctivitis allergic (Eye disorders) | 14
Meibomian gland dysfunction (Eye disorders) | 1
Age-related macular degeneration (Eye disorders) | 1
Corneal erosion (Eye disorders) | 5
Keratitis (Eye disorders) | 1
Corneal disorder (Eye disorders) | 9
Eye pruritus (Eye disorders) | 3
Abnormal sensation in eye (Eye disorders) | 1
Dry eye (Eye disorders) | 12
Eye irritation (Eye disorders) | 22
Ocular hyperaemia (Eye disorders) | 1
Asthenopia (Eye disorders) | 3
Eye pain (Eye disorders) | 4
Eyelids pruritus (Eye disorders) | 1
Blepharitis (Eye disorders) | 8
Eyelid ptosis (Eye disorders) | 1
Blepharal pigmentation (Eye disorders) | 5
Conjunctival erosion (Eye disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 2
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctival deposit (Eye disorders) | 1
Posterior capsule opacification (Eye disorders) | 2
Mydriasis (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 2
Punctate keratitis (Eye disorders) | 14
Diabetic retinopathy (Eye disorders) | 1
Iritis (Eye disorders) | 1
Iris hyperpigmentation (Eye disorders) | 2
Cataract (Eye disorders) | 5
Vision blurred (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Retinal vein occlusion (Eye disorders) | 2
Retinal detachment (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 2
Glaucoma (Eye disorders) | 2
Growth of eyelashes (Eye disorders) | 9
Eyelash thickening (Eye disorders) | 4
Meibomianitis (Eye disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Peripheral artery stenosis (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Intraocular pressure increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.